CLINICAL TRIAL: NCT01319591
Title: Comparison of Creatinine Clearance Calculation Methods for Estimation of Glomerular Filtration Rate in Patients Receiving High-Dose Methotrexate
Brief Title: Comparison of Creatinine Clearance Calculation for Estimation of GFR in Patients Receiving HD Methotrexate
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Audrea Szabatura, Medication Safety Officer, Dana-Farber Cancer Institute
Other Study IDs: 11-043
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: CNS Lymphoma; CNS Involvement of Systemic Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CNS lymphoma patients

SUMMARY:
The purpose of this study is to compare different estimates of calculating creatinine clearance by mathematical formula and compare them to creatinine clearance based on a timed urine collection in patients who received high-dose methotrexate for the treatment of primary CNS lymphoma or CNS involvement of systemic lymphoma.

DETAILED DESCRIPTION:
We intend to perform a retrospective chart review to identify a serum creatinine-based equation that gives the best estimate of CrCl as compared with an equation derived from a 24-hour urine collection.

Study subjects will be identified using the Brigham and Women's Hospital and Dana-Farber Cancer Institute's Adult Pharmacy systems to identify patients who received high-dose methotrexate. Data will be collected starting with December 31, 2010 and proceeding chronologically backwards until the target enrollment of 40 patients is reached.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Received high-dose methotrexate therapy at Dana-Farber Cancer Institute/Brigham and Women's Hospital for the treatment of primary CNS lymphoma or CNS involvement of systemic lymphoma
* Available timed urine collection within 1 week of HDMTX

Exclusion Criteria:

* Receiving high-dose methotrexate for indications other than primary CNS lymphoma or CNS involvement of systemic lymphoma
* Documented viral hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving high-dose methotrexate therapy at Dana-Farber Cancer Institute/Brigham and Women's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
To identify a serum creatinine-based equation that gives the best estimate of CrCl as compared to a measured creatinine clearance formula. | 1 year
  Serum creatinine-based equations to be included in that analysis are: Cockcroft-Gault with the following weight descriptors; ideal body weight, actual body weight, and adjusted body weight; Modified MDRD; CKD-EPI.

SECONDARY OUTCOMES:
To further compare each formula in a different subset of patients. | 1 year
  To further compare each formula in a different subset of patients: Age < 65 years and >/= 65 years; body mass index < 25, 25-30, 30-35, and > 35; serum creatinine <1.5 mg/dL and >/= 1.5 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Audrea H Szabatura, PharmD, BCOP, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No